CLINICAL TRIAL: NCT04377308
Title: Fluoxetine to Reduce Intubation and Death After COVID19 Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Principal Investigator, Cheryl Mccullumsmith, Professor and Chair, Department of Psychiatry, University of Toledo Health Science Campus
Organization: University of Toledo (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FRIDA COVID19
Record Dates: First submitted 2020-04-18; First posted 2020-05-06 (Actual); Results first posted 2022-09-30 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: COVID-19; Cytokine Storm
Keywords: IL-6; fluoxetine; cytokine storm; NF-KB; COVID-19
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome | interventions — Fluoxetine

STUDY DESIGN:
Intervention Model Description: All patients who enter the study will be monitored daily for symptoms of COVID-19. Patients may choose to take fluoxetine or to have treatment as usual. Patients may also choose to have blood drawn and stored for a future analysis of cytokines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment As Usual (No Intervention): Participants may choose to not take fluoxetine and remain in the study
- Fluoxetine (Active Comparator): Participants will take fluoxetine 20 mg initially, increasing as tolerated to a maximum of 60 mg until symptoms abate, then will be tapered by 20 mg per week off the fluoxetine Participants will be on fluoxetine for 2 weeks to 2 months depending on symptom duration
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine — Fluoxetine 20 mg to 60 mg daily given from 2 weeks to 2 months duration
  Other Names: prozac
  Arms: Fluoxetine

SUMMARY:
This project will test the efficacy of fluoxetine to prevent serious consequences of COVID-19 infection, especially death. Becoming sick with COVID-19 virus or any other serious respiratory condition is not fun. However, the dramatic effects of the COVID-19 pandemic on human society stem from its significant mortality, not the number of individuals who become sick. This project aims to prevent serious outcomes such as hospitalization, respiratory failure and death during the time it takes to develop vaccinations and other strategies to prevent COVID-19 infectionPoor outcomes with COVID-19 infection such as hospitalization, respiratory failure, organ failure and death are associated with a dysfunctional exaggerated immune response, called a cytokine storm, that is triggered by Interleukin-6 expression (IL-6) and seems to occur around day 5 to 7 of symptoms. Fluoxetine has extraordinarily strong evidence in its action as a blocker of IL-6 and cytokine storms in both animal models of infection and in human illness such as rheumatoid arthritis and others. This action of fluoxetine is an entirely separate pathway than the serotonergic pathway that allows fluoxetine to act as an antidepressant. This pathway has been demonstrated in cell culture, in animal models, in human illness and by novel bioinformatics analyses of protein transcripts to be relatively unique for fluoxetine and appears to be a novel pathway. This project aims to inhibit the increase in IL-6 expression and thereby prevent the cytokine storm that causes poor outcomes. Patients who have tested positive or are presumptively positive for COVID-19 will be entered into the study and given the option to start the medication fluoxetine, which is demonstrated to prevent IL-6 surges in infectious and inflammatory conditions. Participants will be monitored daily for COVID-19 symptoms and weekly for side effects and tolerance of fluoxetine. A subset of patients will have blood drawn weekly and stored to monitor IL-6 and other cytokine levels at a later date.

This project aims to reduce the serious outcomes of COVID-19 infection by preventing or inhibiting the cytokine storm associated with organ failure, respiratory failure and death.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and above, able to give informed consent or with legally authorized representative
* COVID-19 test positive or presumptive positive awaiting COVID testing or results by following criteria: fever, cough and shortness of breath or presumptive positive by one of these 3 criteria (fever, cough or shortness of breath) and known exposure to COVID-19 positive individual in past 2 weeks

Overall Study Exclusion Criteria :

* Unable to give informed consent and no legal representativ
* Prisoner/ institutionalized patient
* Under age 18

Exclusion from Fluoxetine Arm:

* Active bleeding requiring blood products
* Bipolar disorder not on mood stabilizing medication*
* Known allergy or hypersensitivity to fluoxetine
* Currently taking the following medications : MAO I, pimozide, thioridine
* Currently taking hydroxychloroquine
* Pregnant or breastfeeding
* For hospitalized patients : QTc greater than 500 ms
* *Hospitalized patient may be on hydroxychloroquine if QTc<500 and the primary attending approves

Exclusion from Blood Sample Provision:

* Pregnant
* Self-report of under 110 pounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toledo, Toledo, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment As Usual | Fluoxetine
Started | 4 | 12
Completed | 4 | 11
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment As Usual | Fluoxetine | Total
Number analyzed (Participants) | 4 | 11 | 15
Age, Continuous [Mean (Full Range); unit: Years] | 52 [44 to 61] | 46.09 [24 to 75] | 47.67 [24 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 10 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 11 | 15
Smoke Cigarettes [Count of Participants; unit: Participants]
  Smokes cigarettes | 1 | 1 | 2
  Does not smoke cigarettes | 3 | 10 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Outpatient Subject Hospitalizations
Description: whether the subject is hospitalized for COVID-19 symptoms
Time Frame: 2 months
Population: We had intended this measure for outpatients but had very few study participants who were outpatients.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual | Fluoxetine
Number analyzed (Participants) | 0 | 9
Participants | 0 | 0

2. Primary Outcome: Number of Subjects Undergoing Intubation
Description: whether the subject is intubated for COVID-19 symptoms
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual | Fluoxetine
Number analyzed (Participants) | 4 | 11
Participants | 1 | 0

3. Primary Outcome: Number of Patients Who Died Within 2 Months of Entry Into the Study
Description: Patients who died from any cause within 2 months of entry into the study.
Time Frame: 2 months
Population: review of charts to determine death by any cause within 2 months of entry into study
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual | Fluoxetine
Number analyzed (Participants) | 4 | 11
Participants | 1 | 0

4. Secondary Outcome: Participants With 1 or More Symptom Free Day With no COVID Primary Symptoms During 2 Months After Study Entry
Description: Participant who achieved remission from covid with no active covid symptoms (cough, fever, shortness of breath, fatigue, muscle aches, and loss of taste and smell) from study entry
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual | Fluoxetine
Number analyzed (Participants) | 4 | 11
Participants
  1 or more symptom free days | 3 | 7
  no symptom free days | 1 | 4

5. Secondary Outcome: Participants With Patient Health Questionnaire (PHQ) -9 Score Below 10 After Baseline Assessment
Description: depression score rating from 0 to 27 where higher scores indicate worse depression Scores of 10 or more meet criteria for diagnosis as a mild depressive episode
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual | Fluoxetine
Number analyzed (Participants) | 4 | 10
Participants | 4 | 10

6. Secondary Outcome: Participants With Generalized Anxiety Disorder (GAD) -7 Scale Score Below 10 After Baseline Assessment
Description: anxiety scale with scores ranging from 0 to 21 where higher scores indicate more severe anxiety Scores of 10 or more generally indicate anxiety that might meet criteria for diagnosis as an anxiety disorder
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual | Fluoxetine
Number analyzed (Participants) | 4 | 10
Participants | 4 | 10

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over up to 2 months from when each participant was enrolled by the study team.
Arm/Group | Treatment As Usual | Fluoxetine
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/11
Other Adverse Events (participants affected / at risk) | 0/4 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment As Usual (N=4) | Fluoxetine (N=11)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA — Patient went in to acute respiratory failure secondary to COVID-19 PNA, coded, was emergently intubated and died after attempts to resuscitate. Patient was in the control arm of the study and did not receive the study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT04377308/Prot_SAP_002.pdf